CLINICAL TRIAL: NCT05334784
Title: Use of the Impella ECP in Patients Undergoing an Elective or Urgent High-Risk Percutaneous Coronary Intervention Impella ECP Continued Access Protocol
Brief Title: Impella ECP Study (ECP Study) and Impella ECP Continued Access Protocol
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Abiomed Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABMD-CIP-22-01
Record Dates: First submitted 2022-03-28; First posted 2022-04-19 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: High-Risk Percutaneous Coronary Intervention
Keywords: HRPCI; High-risk percutaneous coronary intervention; Circulatory support; Left ventricular unloading; Abiomed; Impella; Impella ECP; Impella ECP CAP

STUDY DESIGN:
Intervention Model Description: Upon completion of enrollment in the pivotal study, enrollment in Continued Access Protocol will begin.
  ECP Pivotal enrolled 256 subjects and Impella ECP Continued Access Protocol anticipates to enroll up to 600 subjects
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Impella ECP Device (Experimental): Subjects receiving the Impella ECP.
  Interventions: Device: Impella ECP

INTERVENTIONS:
Device: Impella ECP — Subjects will receive the Impella ECP prior to high-risk percutaneous intervention. Device escalation or early termination of the study will be allowed for subjects as deemed necessary by the treating physician. Subjects will be followed until 30-days post-intervention.

SUMMARY:
The Impella ECP Study is a prospective, multi-center, single-arm study evaluating the rate of major adverse cardiovascular and cerebrovascular events (MACCE) with the Impella ECP device in adult patients undergoing elective or urgent high-risk percutaneous coronary intervention.

The above applies to Impella ECP Continued Access Protocol

DETAILED DESCRIPTION:
This is a prospective, multi-center, single-arm study evaluating the major adverse cardiovascular and cerebrovascular event (MACCE) rate of the Impella ECP device in adult patients undergoing elective or urgent high-risk percutaneous coronary intervention (HRPCI). Additionally, this study will evaluate safety related to Impella ECP-related major vascular complications and Impella ECP-related major bleeding. Finally, this study will evaluate secondary endpoints including the occurrence of major hemolysis, aortic valve injury, escalation of care to Impella CP, and the length of hospital stay.

Investigational device products include: Impella ECP pump system (a percutaneous transvalvular micro-axial blood pump), 9Fr introducer sheath, and the automated Impella controller (AIC) with revised console software to allow control of the Impella ECP.

Study flow: Following informed consent, subjects eligible for a HRPCI that meet all of the inclusion and none of the exclusion criteria will be enrolled into the Study. Subjects will undergo Impella ECP placement through a femoral sheath, following crimping of the Impella ECP. The intended coronary intervention will be performed with the mechanical circulatory support provided by the Impella ECP. Once the procedure is completed, the device is weaned and removed. Subjects will be followed for 30 days. Subjects will be treated based on the contemporary AHA/ACC/SCAI practice guidelines throughout the duration of the Study.

A sample size of two hundred seventeen (217) subjects with 30-day follow-up is needed for 90% power at a one-sided 0.05 significance level. Assuming 15% loss-to-follow-up, up to two hundred fifty-six (256) subjects will be enrolled. Safety endpoints will be presented as summary statistics without formal hypothesis testing. The MACCE rate will be assessed against the PG of 24.4% at one-sided 5% significance level.

Impella ECP Continued Access Protocol:

Description, Investigational device and study flow remains the same as above.

A sample size up to six hundred (600) subjects will be enrolled at up to 25 sites. Sites must have been activated in the Pivotal to be eligible for the Continued Access Protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and ≤90 years
2. Subject signed the informed consent
3. Subject is hemodynamically stable and a heart team, including a cardiac surgeon, has determined that an elective or urgent (not emergent) high-risk PCI is the appropriate therapeutic option

Exclusion Criteria:

1. Aortic valve disease that is anticipated to be prohibitive to Impella ECP crossing, including greater than mild aortic stenosis
2. Previous aortic valve replacement or reconstruction
3. Thrombus in left ventricle
4. Subjects with known aortic vessel disease or with aortic dissection
5. Any contraindication that precludes placing an Impella including aortic, iliac or femoral disease such as tortuosity, extensive atherosclerotic disease or stenosis
6. Prior stroke with any permanent, significant (mRS>2), neurologic deficit or any prior intracranial hemorrhage or any prior subdural hematoma or known intracranial pathology pre-disposing to intracranial bleeding, such as an arteriovenous malformation or mass
7. Cardiogenic shock or acutely decompensated pre-existing chronic heart failure. Cardiogenic shock is defined as: systemic hypotension (systolic BP <90 mmHg or the need for inotropes/pressors to maintain a systolic BP >90 mmHg) plus one of the following: any requirement for pressors/inotropes prior to arrival at the catheterization laboratory, clinical evidence of end-organ hypoperfusion or use of IABP or any other circulatory support device
8. Infection of the proposed procedural access site or suspected systemic active infection, including any fever
9. Subject has previously been symptomatic with or hospitalized for COVID-19 unless he/she has been discharged (if hospitalized) and asymptomatic for ≥8 weeks
10. Known contraindication to heparin (i.e., heparin-induced thrombocytopenia), contrast media or Study-required medication(s) (i.e., aspirin)
11. Platelet count <75k, bleeding diathesis, coagulopathy or unwilling to receive blood transfusions
12. Subject is on dialysis
13. Suspected or known pregnancy
14. Subject has other medical, social or psychological problems that, in the opinion of the Investigator, compromises the subject's ability to give written informed consent and/or to comply with study procedures
15. Participation in the active treatment or follow-up phase of another clinical study of an investigational drug or device which has not reached its primary endpoint
16. Subject belongs to a vulnerable population [Vulnerable subject populations are defined as individuals with mental disability, persons in nursing homes, children, impoverished persons, homeless persons, nomads, refugees and those permanently incapable of giving informed consent. Vulnerable populations also may include members of a group with a hierarchical structure such as university students, subordinate hospital and laboratory personnel, employees of the Sponsor, members of the armed forces and persons kept in detention]

The above Inclusion/Exclusion criteria applies for Impella ECP Continued Access Protocol

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 856 (Estimated)
Dates: Start 2022-12-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of MACCE | Device Delivery through 30 Days
  The rate of major adverse cardiovascular and cerebrovascular events (MACCE)
Impella ECP-related major vascular complications (Safety Endpoint 1) | From the Date of Device Delivery through Date of Discharge (assessed up to 30 days)
  Impella ECP-related major vascular complications
Impella ECP-related Major Bleeding (Safety Endpoint 2) | Device Delivery through Discharge from the Index Hospital Admission (assessed up to 30 days)
  Impella ECP-related Major Bleeding

SECONDARY OUTCOMES:
Number of Subjects with Major Hemolysis | Device Delivery through Discharge (assessed up to 30 days)
Number of Subjects with Aortic Valve Injury | Device Delivery through Discharge (assessed up to 30 days)
Number of Subjects with Escalation of Care to Impella CP | Device Removal through Discharge (assessed up to 30 days)
Length of Hospital Stay for enrolled patients | Admission through Discharge (assessed up to 30 days)

CONTACTS AND LOCATIONS:
Overall Officials: Navin Kapur, MD, Study Director — Abiomed Inc.; Seth Bilazarian, MD, Study Director — Abiomed Inc.; Amir Kaki, MD, Principal Investigator — Ascension St. John Hospital
Locations (32):
- United States (32):
  - St. Joseph's Medical Center - Phoenix, Phoenix, Arizona
  - Pima Heart & Vascular, Tucson, Arizona
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Adventist Health Glendale, Glendale, California
  - Keck Hospital of USC, Los Angeles, California
  - Loma Linda University Medical Center, San Bernardino, California
  - Manatee Memorial Hospital, Bradenton, Florida
  - North Florida Regional Medical Center, Gainesville, Florida
  - AdventHealth - Tampa, Tampa, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Ochsner Foundation Hospital, New Orleans, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Ascension St. John Hospital, Detroit, Michigan
  - Spectrum Health, Grand Rapids, Michigan
  - St. Cloud (CentraCare), Saint Cloud, Minnesota
  - Providence St. Patrick, Missoula, Montana
  - Hackensack University Medical Ctr, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - The Valley Hospital, Ridgewood, New Jersey
  - New Mexico Heart Institute, Albuquerque, New Mexico
  - Buffalo General, Buffalo, New York
  - CUMC/ New York Presbyterian Hospital, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Oklahoma Heart Hospital - South, Oklahoma City, Oklahoma
  - Providence St. Vincent Med Center, Portland, Oregon
  - TriStar Centennial Medical Center, Nashville, Tennessee
  - Texas Health Presbyterian Hospital Dallas, Dallas, Texas
  - Baylor Scott & White The Heart Hospital Plano, Plano, Texas
  - Methodist Hospital - San Antonio, San Antonio, Texas
  - Sentara Norfolk Health System, Norfolk, Virginia
  - West Virginia University Hospital, Morgantown, West Virginia